CLINICAL TRIAL: NCT02887235
Title: Food as Medicine: A Phase III Randomized Controlled Trial of Home Delivered, Medically Tailored Meals (HDMTM) on Quality of Life in Metastatic Lung and Non-colorectal GI Cancer Patients
Brief Title: Food as Medicine: An RCT to Study the Effect of Home Delivered, Medically Tailored Meals on Patients With Metastatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: s15-00708
Record Dates: First submitted 2016-08-08; First posted 2016-09-02 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SOC) Meals (No Intervention): Patient assigned in this arm will receive standard of care nutritional services including nutrition consult, evaluation, and as needed follow-ups.
- Medically tailored meals (Active Comparator): Patient assigned in this arm will receive home delivered, medically tailored meals (HDMTM) in addition to the standard nutritional care.
  Interventions: Other: Home Delivered, Medically Tailored Meals (HDTM)

INTERVENTIONS:
Other: Home Delivered, Medically Tailored Meals (HDTM)
  Arms: Medically tailored meals

SUMMARY:
The purpose of this study is to determine whether medically tailored meals (HDTM) can improve quality of life for patients with metastatic cancer.

DETAILED DESCRIPTION:
The current standard of care at the cancer center is for all patients receiving cytotoxic therapy to undergo a nutritional consultation and evaluation with a registered oncology dietitian. The goal of this consultation is to prevent nutritional deficiencies, promote optimal nutritional intake, hydration, and weight maintenance, as well as maintain lean body mass.

All patients on this study will receive standard of care nutritional services including nutrition consult, evaluation, and as needed follow-ups. However, patients randomized to arm 2 will receive home delivered, medically tailored meals in addition to the standard nutritional care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pathologically confirmed metastatic pancreatic, hepatobiliary, esophageal, or lung cancer, either newly metastatic or metastatic at presentation (M1+) and enrollment within 6 weeks of diagnosis; measurable disease need not be present.
* Pain Score (PS) 0-3
* Age>18
* Both male and female subjects eligible
* All ethnicities eligible
* Access to refrigerator or freezer

Exclusion Criteria:

* Diagnosis of metastatic cancer no greater than 6 weeks prior to expected study enrollment
* Currently receiving home delivered meals from other sources
* Evidence of any alimentary tract obstruction or other condition preventing oral alimentation
* Requirement for enteral or parenteral nutrition at time of diagnosis
* Incarcerated individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Quality of life measurement | At 12 weeks follow up
  Quality of life will be assessed using the Functional Assessment in Cancer Therapy - General (FACT-G). Developed by Cella et al. the FACT-G is a well validated and widely used multi-dimensional health related quality of life measure for cancer patients. It consists of 28 self-assessment items on a 5 point Likert scale that address four domains:
  physical well-being, social/family well-being, emotional well-being, and functional well-being. Scores are calculated for each sub-scale per FACT scoring instructions and summed for a total score ranging between 0 and 108 with higher scores indicating a higher quality of life.

SECONDARY OUTCOMES:
Change in mood assessment | From baseline to 12 weeks
  The Hospital Anxiety Depression Survey will be utilized to assess patient mood on this study. It is a validated, 14 item self-assessment tool used to assess severity of anxiety and depression symptoms in patients. Two 7 item subscales assess anxiety and depression in the past one week. Item responses are integer values between 0-3 and values for each subscale are added to give a subscale score. Scores on each subscale can range from 0 to 21 and a score greater than 11 is considered consistent with anxiety or depression. Scores of 7 or less are considered normal and scores of 8 to 10 are borderline. A score of 8 or greater on the anxiety subscale has a sensitivity of 0.9 and specificity of 0.78 for anxiety. Similarly, a score of 8 or greater on the depression subscale has a sensitivity of 0.83 and specificity of 0.79 for depression.
Patient weight assessment | From baseline to 12 weeks
  Weight is measured at each physician visit per hospital policy. Weight at each interval will be recorded in the electronic medical record (EMR). Should the patient not have a scheduled visit with their primary oncologist or registered dietitian within the required visit window, any weight recorded in the EMR within the visit window can be used. The changes in weight from baseline to 12 weeks,will be measured using the Abridged Patient Generated Subjective Global Assessment (abPG-SGA) in the 2 arms.
Nutritional status assessment | From baseline to 12 weeks
  The change in nutritional status from baseline will be measured using the Abridged Patient Generated Subjective Global Assessment (abPG-SGA) in the 2 arms.
Financial toxicity assessment | From baseline to 12 weeks
  In 2014 a novel instrument to assess subjective financial toxicity, the Financial Toxicity Patient-Reported Outcome in Cancer measure (COST) was designed and recently validated. It is an 11 item assessment with 5 point Likert scale responses developed by de Souza et al reference to assess the levels of financial distress experienced by cancer patients. Each item response is scored 0-4 and then all individual item scores are summed. For incomplete surveys, the sum score is multiplied by 11 and then divided by the number of items answered. Total scores can range from 0-44 with higher scores representing higher subjective patient financial toxicity.
Food security assessment plus HDMTM from baseline to 12 weeks | From baseline to 12 weeks
  U.S. Adult Food Security Survey module to assess food security.It is a 10 item questionnaire developed by the US Department of Agriculture to specifically assess food insecurity in adults. Affirmative responses to each item are given one point. Total raw scores are calculated by adding all points (affirmative responses) and can range from 0-10. A raw score of zero is considered high food security. A raw score 1-2 is considered marginal food security. A raw score 3-5 is considered low food security and raw scores 6-10 are very low food security.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schiff, MD, PhD, Principal Investigator — NYU Perlmutter Cancer Center
Locations (1):
- NYU Perlmutter Cancer Center, New York, New York, United States